CLINICAL TRIAL: NCT00758940
Title: A Six-months, Open-labelled Clinical Assessment of Visual Function After Bilateral Implantation of Arcysof ReSTOR Multifocal Intra-ocular Lens
Brief Title: Clinical Assessment of Visual Function With the Acrysof ReSTOR Multifocal IOL
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary Investigator resigned from Hospital
Sponsor: Alcon Research (Industry)
Responsible Party: Ricky Ho, RA Manager, Alcon Research Ltd.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HK-Restor-YIU-01
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2010-01

CONDITIONS: Visual Outcomes
Keywords: Clinical; assessment; of visual; function; with the Acrysof ReSTOR; multifocal IOL

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Acrysof ReSTOR multifocal IOL
  Interventions: Device: Acrysof ReSTOR multifocal IOL

INTERVENTIONS:
Device: Acrysof ReSTOR multifocal IOL — Implanted into the study eye following cataract extraction surgery

SUMMARY:
An unmasked trial after bilateral implantation of AcrySof® ReSTOR®, SA60D3 IOL . Enrolled are at least 30 patients or as much as possible from the doctor's clinical practice perspective. 6 months follow-up after IOL implant in the 2nd eye

ELIGIBILITY:
Inclusion Criteria:

* Able to complete all required postoperative visits; Planned cataract removal by phaco; 21 years of age or older, either gender or any race; potential postoperative visual acuity of 20/20; astigmatism ≦1.0D measured by keratometry in study eye(s);clear int

Exclusion Criteria:

* Signs of capsular tear, significant anterior chamber hyphema;zonular rupture; corneal pathology and refractive surgery;hypercritical patient; patients with unrealistic expectations in post-op VA; happy to wear glasses;occupational night drivers

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Near,intermediate,distance visual acuity | pre-op;1 week after 1st eye surgery,1month and 6 month after 2nd eye surgery

SECONDARY OUTCOMES:
contrast sensitivity | 6 month after 2nd eye surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States